CLINICAL TRIAL: NCT00363766
Title: A Phase 2 Study of LY573636-Sodium Administered as an Intravenous Infusion on Day 1 of a 21-Day Cycle as Third-line Treatment in Patients With Unresectable, Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of LY573636-Sodium in Patients With Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9813; H8K-MC-JZAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

ARMS (1):
- LY573636 (Experimental)
  Interventions: Drug: LY573636-sodium

INTERVENTIONS:
Drug: LY573636-sodium — A loading dose to target 420 micrograms/milliliter (µg/mL) maximum concentration (Cmax) or 380 µg/mL Cmax followed by a lower chronic dose to maintain Cmax within these target ranges, intravenous, every 21 days until disease progression.
  Other Names: Tasisulam

SUMMARY:
The primary objective is to estimate the time to progressive disease for patients who receive LY573636-sodium (hereafter referred to as LY573636) after two previous treatments for metastatic non-small cell lung cancer. Patients will receive an intravenous infusion of study drug once every 21 days. Computed tomography (CT)-scans will be done before the first dose and then after every other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic non-small-cell lung cancer
* At least 18 years of age
* Have received 2 previous treatment regimens for metastatic non-small-cell lung cancer

Exclusion Criteria:

* Serious pre-existing medical conditions
* Previous cancer (except skin cancer, excluding melanoma)
* Have received 3 or more previous treatment regimens for metastatic non- small-cell lung cancer
* Active treatment with Coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gauting
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Löwenstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sisto

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LY573636 Target Cmax 420 µg/mL: A loading dose of LY573636 to target 420 micrograms/milliliter (µg/mL) maximum concentration (Cmax) followed by a lower chronic dose to maintain Cmax within this target range, intravenous, every 21 days until disease progression.
- LY573636 Target Cmax 380 µg/mL: A loading dose of LY573636 to target 380 µg/mL Cmax followed by a lower chronic dose to maintain Cmax within this target range, intravenous, every 21 days until disease progression.
Period: Overall Study
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Started | 32 | 20
Completed | 0 | 0
Not Completed | 32 | 20
Not completed — Progressive Disease | 15 | 9
Not completed — Adverse Event | 10 | 2
Not completed — Disease Related Death | 1 | 3
Not completed — Not Disease Related Death | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL | Total
Number analyzed (Participants) | 32 | 20 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.14) | 61.1 (7.90) | 60.2 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 25 | 14 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 32 | 20 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 19 | 11 | 30
  Italy | 13 | 9 | 22
Pathological Diagnosis [Count of Participants; unit: Participants]
  Lung, Large Cell | 2 | 0 | 2
  Poorly Differentiated Non-Small-Cell Lung Cancer | 6 | 1 | 7
  Lung, Adenocarcinoma | 12 | 12 | 24
  Lung, Squamous Cell | 11 | 7 | 18
  Bronchoalveolar Carcinoma | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death from study disease. PD was determined using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.0). PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: First dose to measured progressive disease or death from study disease up to 10.35 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 32 | 20
months | 3.12 [2.04 to 4.21] | 1.64 [1.35 to 5.19]

2. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.0). PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: First treatment dose to measured progressive disease or death from any cause up to 10.35 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- LY573636 Target Cmax 380 µg/mL: A loading of LY573636 dose to target 380 µg/mL Cmax followed by a lower chronic dose to maintain Cmax within this target range, intravenous, every 21 days until disease progression.
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 32 | 20
months | 2.69 [1.38 to 4.17] | 1.43 [1.31 to 3.22]

3. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Objective Response Rate)
Description: Objective response rate is the percentage of participants with complete response (CR) + partial response (PR), as assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.0). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: First treatment dose to measured progressive disease or death due to any cause up to 10.35 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 32 | 20
percentage of participants | 0 | 0

4. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY573636
Time Frame: Predose up to 2 hours postdose in Cycles 1 and 2 (21 days cycle)
Population: Participants who received study drug and had pharmacokinetic (PK) data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 25 | 20
micrograms/milliliter (µg/mL)
  Cycle 1 | 379.6 (14.1) | 337.6 (15.5)
  Cycle 2: number analyzed (Participants) | 13 | 12
  Cycle 2 | 293.7 (11.0) | 316.1 (14.4)

5. Secondary Outcome: Overall Survival Time
Description: Defined as the time from date of first dose to the date of death due to any cause.
Time Frame: First treatment dose to death due to any cause up to 25.23 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 32 | 20
months | 8.48 [5.06 to 10.15] | 7.97 [4.07 to 12.06]

6. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression of disease or death due to any cause. CR or PR is classified according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines (version 1.0). CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Time of response to progressive disease or death up to 10.35 months
Population: Since there were zero participants with CR or PR, the duration of response could not be analyzed.
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease (SD) is defined from date of documented SD or better to first date of progression of disease (PD) (assessed every cycle during study therapy, or every 2 months during post-therapy until PD). SD is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for PD. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Time from documented stable disease or better to first date of progressive disease up to 10.35 months
Population: All enrolled participants who received at least 1 dose of study drug and had a best overall response of stable disease or better.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 14 | 7
months | 4.21 [3.58 to 5.72] | 4.93 [3.22 to 10.35]

8. Secondary Outcome: Number of Participants With Adverse Events (Safety)
Description: Data are presented as number of participants who experienced serious adverse events or all other nonserious adverse events during the study. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Event section.
Time Frame: First treatment dose up to 25.23 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Number analyzed (Participants) | 32 | 20
Participants
  Serious Adverse Events | 17 | 9
  Other Nonserious Adverse Events | 30 | 17

ADVERSE EVENTS:
Arm/Group | LY573636 Target Cmax 420 µg/mL | LY573636 Target Cmax 380 µg/mL
Serious Adverse Events (participants affected / at risk) | 17/32 | 9/20
Other Adverse Events (participants affected / at risk) | 30/32 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636 Target Cmax 420 µg/mL (N=32) | LY573636 Target Cmax 380 µg/mL (N=20)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (11) | 2 (2)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Condition Aggravated (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0)
Superior Vena Caval Occlusion (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636 Target Cmax 420 µg/mL (N=32) | LY573636 Target Cmax 380 µg/mL (N=20)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (11) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 4 (6) | 1 (1)
Face Oedema (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 11 (11) | 7 (7)
General Physical Health Deterioration (General disorders) | 2 (2) | 0 (0)
Mucosal Inflammation (General disorders) | 2 (3) | 2 (2)
Oedema Peripheral (General disorders) | 5 (8) | 2 (2)
Pyrexia (General disorders) | 6 (8) | 2 (2)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 2 (2) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (2)
Forced Expiratory Volume (Investigations) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil Count (Investigations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Neuropathy Peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 3 (3) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Embolism (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days